CLINICAL TRIAL: NCT02264210
Title: A Randomized, Phase II Trial of Icotinib Versus Observation as Adjuvant Treatment in Stage IB Non-Small Cell Lung Cancer Harboring Activating Epidermal Growth Factor Receptor Mutation
Brief Title: Icotinib for Completed Resected IB NSCLC With EGFR Mutation
Acronym: CORIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1003; wsy004 (Other: Guangdong Province Association Study of Thoracic Oncology)
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Lung Neoplasms; Squamous Cell Lung Cancer; Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Large Cell Lung Cancer; Bronchial Neoplasms; Stage IB Non-small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Bronchial Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Icotinib 125 mg three times daily (375 mg per day) orally for 12 months.
  Interventions: Drug: Icotinib
- Observation group (No Intervention): Observation.

INTERVENTIONS:
Drug: Icotinib — Icotinib 125 mg three times daily (375 mg per day) by mouth for 12 months.
  Other Names: BPI-2009; Conmana
  Arms: Intervention group

SUMMARY:
This phase II trial studies how well icotinib works in treating patients with completely resected stage IB NSCLC harboring EGFR mutation.

DETAILED DESCRIPTION:
Adjuvant chemotherapy have shown little evidence of survival benefit in patients with stages IB non-small cell lung cancer (NSCLC) after complete resection. Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) show great efficacy in patients with EGFR mutant non-small cell lung cancer (NSCLC). Icotinib is a novel EGFR-TKI developed by a group of Chinese scientists and clinician. In the phase III ICOGEN trial, icotinib had non-inferiority efficacy to gefitinib with better safety. This study is studying icotinib to see how well it works in treating patients with fully resected stage IB NSCLC harboring EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males or females, Aged 18-75 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Had completely resected pathological confirmed stage IIA-IIIA NSCLC.
* EGFR activating mutation in exon 19 or 21.
* Patient who can start the investigational therapy within 3-6 weeks after the complete resection.
* ECOG performance status of 0-1.
* Had a life expectancy of 12 weeks or more.
* Adequate hematological function, adequate liver function and renal function.
* Female patients, except those who are postmenopausal or surgically sterilized, must have a negative pre-study serum or urine pregnancy test.

Exclusion Criteria:

* Had had previous chemotherapy, radiotherapy, or agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Inability to comply with protocol or study procedures.
* Had a history another malignancy in the last 5 years with the exception of cured basal cell carcinoma of the skin, cured in situ carcinoma of the uterine cervix and cured epithelial carcinoma of the bladder.
* Any evidence confirmed tumor recurrence before investigational therapy.
* Known severe hypersensitivity to icotinib or any of the excipients of this product.
* Evidence of clinically active interstitial lung disease.
* Eye inflammation not fully controlled or conditions predisposing the subject to this.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Known human immunodeficiency virus (HIV) infection.
* Pregnancy or breast-feeding women.
* Ingredients mixed with small cell lung cancer patients.
* History of neurologic or psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, MD, Principal Investigator — Guangdong Province Association Study of Thoracic Oncology
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ou W, Li N, Wang BX, Zhu TF, Shen ZL, Wang T, Chang WG, Chang ZH, Hu XX, Pu Y, Ding LM, Wang SY. Adjuvant icotinib versus observation in patients with completely resected EGFR-mutated stage IB NSCLC (GASTO1003, CORIN): a randomised, open-label, phase 2 trial. EClinicalMedicine. 2023 Feb 3;57:101839. doi: 10.1016/j.eclinm.2023.101839. eCollection 2023 Mar. PMID 36816343

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Observation Group
Started | 63 | 65
Completed | 63 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Observation Group: Observation only group.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Observation Group | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Continuous [Median (Full Range); unit: Years] | 56 [35 to 75] | 57 [32 to 75] | 56 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 26 | 27 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 63 | 65 | 128
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
EGFR mutation site [Count of Participants; unit: Participants]
  Exon 19 deletion | 32 | 30 | 62
  Exon 21 L858R | 29 | 34 | 63
  Exon 18 G719X | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: 3-year Disease-Free Survival
Description: 3-year DFS was defined as the percentage of patients who were disease free at 3 years. 3-year DFS were calculated by the Kaplan-Meier method, and the difference in 3-year DFS between groups was compared by the Z test.
Time Frame: From randomization to the time of disease recurrence or death as a result of any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: Percentage of patients at 3 years
Groups:
- Observation Group: Observation alone group.
Arm/Group | Intervention Group | Observation Group
Number analyzed (Participants) | 63 | 65
Percentage of patients at 3 years | 96.1 [91.3 to 99.9] | 84.0 [75.1 to 92.9]

ADVERSE EVENTS:
Time Frame: 1 year
Description: All AEs were classified according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0.
Arm/Group | Intervention Group | Observation Group
All-Cause Mortality (participants affected / at risk) | 0/63 | 3/65
Serious Adverse Events (participants affected / at risk) | 4/63 | 0/65
Other Adverse Events (participants affected / at risk) | 49/63 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=63) | Observation Group (N=65)
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=63) | Observation Group (N=65)
Rash (Skin and subcutaneous tissue disorders) | 25 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 0
Pain (General disorders) | 7 | 0
Elevated ALT (Blood and lymphatic system disorders) | 6 | 0
Decreased appetite (General disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT02264210/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT02264210/SAP_001.pdf